CLINICAL TRIAL: NCT00475904
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled Non-inferiority Trial of EpiCept™ NP-1 Topical Cream (2% Ketamine / 4% Amitriptyline) vs. Oral Gabapentin in Postherpetic Neuralgia (PHN)
Brief Title: A Comparison of EpiCept™ NP-1 Topical Cream vs. Oral Gabapentin in Postherpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EpiCept Corporation (Industry)
Responsible Party: Stephane Allard, Chief Medical Officer, EpiCept Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPC2007-02
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Post Herpetic Neuralgia; PHN; Neuropathy; Nerve Pain
Keywords: Post Herpetic Neuralgia; PHN; Neuropathy; Nerve Pain; Topical
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- amitriptyline 4% ketamine 2% cream, placebo capsules (Active Comparator): Np-1 cream and placebo gabapentin
  Interventions: Drug: EpiCept-NP-1 Cream
- gabapentin capsules, placebo cream (Active Comparator): gabapentin caps and placebo cream
  Interventions: Drug: Gabapentin Capsules
- placebo cream and capsules (Placebo Comparator): placebo cream and capsules
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: EpiCept-NP-1 Cream — ketamine 4% amitriptyline 2% cream, twice daily for 4 weeks
  Arms: amitriptyline 4% ketamine 2% cream, placebo capsules
Drug: Gabapentin Capsules — 1800mg/day capsules for 4 weeks
  Other Names: gabapentin, neurontin
  Arms: gabapentin capsules, placebo cream
Drug: placebo — placebo cream and caps
  Other Names: vehicle cream, placebo capsules
  Arms: placebo cream and capsules

SUMMARY:
The purpose of this study is to compare EpiCept™ NP-1 Topical Cream (2% ketamine / 4% amitriptyline) vs. Oral Gabapentin in the treatment of Postherpetic Neuralgia (PHN)

DETAILED DESCRIPTION:
This is a phase II, multicenter, double-blind, randomized, placebo-controlled, parallel group study of NP-1 and oral gabapentin in approximately 500 patients with PHN. Adult patients with pain resulting from PHN and meeting all other eligibility requirements will be screened for 7 days to determine their average daily pain intensity. Qualifying patients will be randomized on a 2:2:1 basis to NP-1, oral gabapentin, or placebo. The treatment period will be 4-Weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with pain for ≥ 3 months following onset of a herpes zoster rash

Exclusion Criteria:

* Clinically significant intercurrent illness (e.g., endocrine, cardiac, hepatic, renal, neurologic, hematologic, skeletal) that the investigator determines could interfere with the efficacy or safety assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Dworkin, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- Multiple Centers, New Delhi, India

RESULTS

PARTICIPANT FLOW:
Groups:
- Amitriptyline 4% Ketamine 2% Cream, Placebo Capsules: amitriptyline 4% ketamine 2% cream 4grams applied twice daily to affected area, placebo capsules taken orally 3 times daily
- Gabapentin Capsules, Placebo Cream: oral gabapentin capsules 600mg three times daily and placebo cream applied 4 grams twice daily
- Placebo Cream and Capsules: placebo NP-1 cream 4gms applied twice daily and placebo gabapentin capsules, taken orally 3 times daily
Period: Overall Study
Arm/Group | Amitriptyline 4% Ketamine 2% Cream, Placebo Capsules | Gabapentin Capsules, Placebo Cream | Placebo Cream and Capsules
Started | 140 | 144 | 76
Completed | 125 | 131 | 72
Not Completed | 15 | 13 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amitriptyline 4% Ketamine 2% Cream, Placebo Capsules | Gabapentin Capsules, Placebo Cream | Placebo Cream and Capsules | Total
Number analyzed (Participants) | 140 | 144 | 76 | 360
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 106 | 109 | 55 | 270
  >=65 years | 34 | 35 | 21 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 51.3 (16.04) | 53.2 (15.53) | 53.2 (16.47) | 52.5 (15.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 49 | 30 | 135
  Male | 84 | 95 | 46 | 225
Region of Enrollment [Number; unit: participants]
  India | 140 | 144 | 76 | 360

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scores Comparing NP-1 Cream vs. Placebo Cream for Treatment of the Pain of Post Herpetic Neuralgia(PHN)From Baseline to 28 Days.
Description: Difference in pain scores between NP-1 cream vs. placebo cream for the treatment of the pain of PHN. Baseline pain scores were compared to the pain scores after 28 days of treatment. Pain scores were rated on a 11 point numerical rating scale (0-10) where 0 was no pain and 10 was worst possible pain.
Time Frame: baseline and 28 days
Population: This analysis was performed for the Intent To Treat (ITT) population using the ast Observation Carried Forward (LOCF) approach.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Amitriptyline 4% Ketamine 2% Cream, Placebo Capsules | Gabapentin Capsules, Placebo Cream | Placebo Cream and Capsules
Number analyzed (Participants) | 135 | 138 | 76
units on a scale | 2.424 [2.07 to 2.78] | 2.471 [2.17 to 2.77] | 1.877 [1.43 to 2.32]
Statistical Analysis 1: Comparison: Amitriptyline 4% Ketamine 2% Cream, Placebo Capsules vs Placebo Cream and Capsules; In the initial analysis, the efficacy of the test treatment NP-1 cream was compared with placebo using an analysis of variance (ANOVA). The analysis was conducted using the ITT population to compare the mean changes in pain scores from baseline to endpoint for the 2 treatments; the LOCF approach was employed for patients who did not complete the trial; Test type: Superiority or Other; p = 0.0441, ANOVA — a priori threshold for statistical significance was p<0.05; Mean Difference (Final Values) = 0.547, 95% CI 2-sided [0.01 to 1.08], Standard Error of Mean 0.2709

2. Primary Outcome: Change in Pain Intensity From Baseline to 28 Days of Treatment, Comparison Between NP-1 Topical Cream and Oral Gabapentin
Description: Change in pain intensity scores between NP-1 cream vs. oral gabapentin for the treatment of the pain of PHN. Baseline pain scores were compared to the pain scores after 28 days of treatment. Pain scores were rated on a 11 point numerical rating scale (0-10) where 0 was no pain and 10 was worst possible pain.
Time Frame: baseline to 28 Days
Population: Intent To Treat (ITT) population using the Last Observation Carried Forward) LOCF imputation technique
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Amitriptyline 4% Ketamine 2% Cream, Placebo Capsules | Gabapentin Capsules, Placebo Cream | Placebo Cream and Capsules
Number analyzed (Participants) | 135 | 138 | 76
units on a scale | 2.424 [2.07 to 2.7] | 2.471 [2.17 to 2.77] | 1.877 [1.43 to 2.3]
Statistical Analysis 1: Comparison: Amitriptyline 4% Ketamine 2% Cream, Placebo Capsules vs Gabapentin Capsules, Placebo Cream; the primary hypothesis of this study was that NP-1 topical cream (amitriptyline 4%/ketamine 2%) administered twice daily in doses of 4 gm for 4 weeks is not inferior to the standard treatment (oral gabapentin 600 mg 3 times daily) for relieving the pain of adult patients with PHN; Test type: Non-Inferiority or Equivalence — To conclude that the NP-1 was not inferior to gabapentin, the upper limit of the 2-sided 90% CI for the difference between treatments for the endpoint mean pain score was required to be below the non-inferiority margin of 0.70; p = 0.8409, ANCOVA — To conclude that the NP-1 was not inferior to gabapentin, the upper limit of the 2-sided 90% CI for the difference between treatments for the endpoint mean pain score was required to be below the non-inferiority margin of 0.70; Mean Difference (Final Values) = 0.046, 90% CI 2-sided [-0.33 to 0.43], Standard Error of Mean .2311

ADVERSE EVENTS:
Arm/Group | Amitriptyline 4% Ketamine 2% Cream, Placebo Capsules | Gabapentin Capsules, Placebo Cream | Placebo Cream and Capsules
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/144 | 0/76
Other Adverse Events (participants affected / at risk) | 7/140 | 2/144 | 1/76
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amitriptyline 4% Ketamine 2% Cream, Placebo Capsules (N=140) | Gabapentin Capsules, Placebo Cream (N=144) | Placebo Cream and Capsules (N=76)
Vertigo (Ear and labyrinth disorders) | 7 (7) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No